CLINICAL TRIAL: NCT05499260
Title: A Randomized, Double-blind, Placebo-controlled, Phase I Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of Single and Multiple Ascending Oral Doses of CB03-154 in Healthy Subjects.
Brief Title: A Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of CB03-154 in Healthy Participants
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Zhimeng Biopharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CB03-154-101
Record Dates: First submitted 2022-08-08; First posted 2022-08-12 (Actual); Last update posted 2022-08-16 (Actual); Status verified 2022-08

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (17):
- CB03-154 SAD 5mg (Experimental): Participants will receive CB03-154 5mg orally once daily in a fasted state.
  Interventions: Drug: CB03-154
- Placebo SAD 5mg (Placebo Comparator): Participants will receive placebo 5mg orally once daily in a fasted state.
  Interventions: Drug: Placebo
- CB03-154 SAD 10mg (Experimental): Participants will receive CB03-154 10mg orally once daily in a fasted state.
  Interventions: Drug: CB03-154
- Placebo SAD 10mg (Placebo Comparator): Participants will receive placebo 10mg orally once daily in a fasted state.
  Interventions: Drug: Placebo
- CB03-154 SAD 20mg (Experimental): Participants will receive CB03-154 20mg orally once daily in a fasted state.
  Interventions: Drug: CB03-154
- Placebo SAD 20mg (Placebo Comparator): Participants will receive placebo 20mg orally once daily in a fasted state.
  Interventions: Drug: Placebo
- CB03-154 SAD 40mg (Experimental): Participants will receive CB03-154 40mg orally once daily in a fasted state.
  Interventions: Drug: CB03-154
- Placebo SAD 40mg (Placebo Comparator): Participants will receive placebo 40mg orally once daily in a fasted state
  Interventions: Drug: Placebo
- CB03-154 SAD 60mg (Experimental): Participants will receive CB03-154 60mg orally once daily in a fasted state.
  Interventions: Drug: CB03-154
- Placebo SAD 60mg (Placebo Comparator): Participants will receive placebo 60mg orally once daily in a fasted state.
  Interventions: Drug: Placebo
- CB03-154 FE (Experimental): Participants will receive CB03-154 orally once daily in a fed state.
  Interventions: Drug: CB03-154
- CB03-154 MAD 10mg (Experimental): Participants will receive CB03-154 10mg orally once daily in a fasted state, for 14 consecutive days.
  Interventions: Drug: CB03-154
- Placebo MAD 10mg (Placebo Comparator): Participants will receive placebo 10mg orally once daily in a fasted state, for 14 consecutive days.
  Interventions: Drug: Placebo
- CB03-154 MAD 20mg (Experimental): Participants will receive CB03-154 20mg orally once daily in a fasted state, for 14 consecutive days.
  Interventions: Drug: CB03-154
- Placebo MAD 20mg (Placebo Comparator): Participants will receive placebo 20mg orally once daily in a fasted state, for 14 consecutive days.
  Interventions: Drug: Placebo
- CB03-154 MAD 40mg (Experimental): Participants will receive CB03-154 40mg orally once daily in a fasted state, for 14 consecutive days.
  Interventions: Drug: CB03-154
- Placebo MAD 40mg (Placebo Comparator): Participants will receive placebo 40mg orally once daily in a fasted state, for 14 consecutive days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CB03-154 — CB03-154 tablet once daily.
  Arms: CB03-154 FE; CB03-154 MAD 10mg; CB03-154 MAD 20mg; CB03-154 MAD 40mg; CB03-154 SAD 10mg; CB03-154 SAD 20mg; CB03-154 SAD 40mg; CB03-154 SAD 5mg; CB03-154 SAD 60mg
Drug: Placebo — Placebo tablet once daily.
  Arms: Placebo MAD 10mg; Placebo MAD 20mg; Placebo MAD 40mg; Placebo SAD 10mg; Placebo SAD 20mg; Placebo SAD 40mg; Placebo SAD 5mg; Placebo SAD 60mg

SUMMARY:
CB03-154 is an investigational drug developed by Shanghai Zhimeng Biopharma Inc. for the treatment of Epilepsy.

DETAILED DESCRIPTION:
The purpose of this study is to see how safe the study drug is and how well it is tolerated after dosing. The study will also test how the study drug is taken up and eliminated by the body. An additional part of the study is to look at how this could be changed by giving the study drug with food.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female 18 to 55 years of age, inclusive.
2. Ability to understand and willingness to sign a written informed consent form.
3. Healthy as determined by medical history, physical examination, laboratory parameters, vital signs, and ECG at Screening and Check-in.
4. Body mass index (BMI) ≥18.0 to ≤32.0 kg/m2 and body weight >50 kg (males) or >45 kg (females) at Screening.
5. If a female, must be:

   * Postmenopausal, defined as amenorrhea for at least 12 months, and confirmed by serum follicle stimulating hormone (FSH) and estradiol levels at Screening, OR
   * Surgically sterile with a documented hysterectomy, partial hysterectomy, bilateral oophorectomy, or bilateral tubal ligation at least 6 months prior to Screening, OR
   * If of child-bearing potential, sexually active females with male partners must be using an acceptable method of contraception such as an intrauterine device, implant or contraceptive injection, or two forms of the following (e.g., diaphragm, cervical cap, oral, patch or vaginal hormonal contraceptive, condom, spermicide, or sponge) for the last three months, and agree to continue to use their method of birth control for the duration of the study and for a minimum of one complete menstrual cycle after study completion. If a female subject is abstinent, she must agree to use an acceptable form of birth control should she become sexually active during the study.
6. If a female, must have a negative pregnancy test result at Screening and Check-in.
7. If a male, if sexually active with a female partner of child-bearing potential and has not had a vasectomy, must agree to use a highly effective double barrier method of contraception as deemed appropriate by the Investigator and must not donate sperm during the study and for 3 months after the last dose of study drug.
8. Non-smokers (including nicotine-containing products) for at least 6 continuous months prior to the first dose by subject report.
9. Willingness and ability to comply with study procedures and follow-up examination.

Exclusion Criteria:

1. Reported history of or current clinically significant medical illness including but not limited to cardiac, hepatic, renal, respiratory, gastrointestinal, endocrine, immunologic, dermatologic, hematologic, neurological (e.g. history of epileptic seizures), or psychiatric disease.
2. Reported history or presence of pro-arrhythmic conditions, including a marked baseline prolongation of QTc interval (i.e., repeated demonstration of a QTcF interval >450 milliseconds) or a history of additional significant risk factors for torsade de pointes (e.g., family history of long QT syndrome), including any evidence of QTcF prolongation at screening.
3. Clinically significant abnormal values for hematology, clinical chemistry, or urinalysis at Screening or Check-in as deemed by the Investigator.
4. Systolic blood pressure > 140 mm Hg and/or diastolic blood pressure > 90 mm Hg at Screening, and determined by the Investigator to confer a safety risk to the subject. Blood pressure measurements may be repeated after at least 10 minutes of rest if initial values obtained at Screening or Check-in are exclusionary.
5. Subjects with active pathogen infections or carrier including but not limited to testing positive at Screening for human immunodeficiency virus (HIV), Hepatitis B surface antigen (HBsAg), or Hepatitis C virus (HCV) antibody.
6. Subjects with a positive test result for Coronavirus disease 2019 (COVID-19) at Check-in.
7. Donated blood or blood product or had substantial loss of blood (more than 500 mL) within 3 months prior to Screening.
8. Use of any prescription or non-prescription drugs (including vitamins and herbal supplements) within 7 days prior to the first dose of study drug and throughout the study. Use of the following medication will be allowed during the study: acetaminophen (up to 1000 mg per 24 hours at the discretion of the Investigator).
9. Reported history and/or recent evidence (within 2 years prior to the Screening) of alcohol abuse (e.g., for females, 4 or more drinks during a single occasion, or 8 or more drinks per week, and for males, 5 or more drinks during a single occasion, or 15 or more drinks per week), or other drug/substance use disorder.
10. Positive test result for alcohol and/or drugs of abuse at Screening or Check-in.
11. Known allergy or hypersensitivity to CB03-154 or any of excipients of CB03-154 tablet formulation.
12. Received an experimental drug or used experimental medical device within 3 months or within 10 half-lives of the drug, whichever is longer, prior to the first dose of study drug.
13. Any condition or disorder that in the Investigators' opinion would put the subject or study conduct at risk if the subject were to participate in the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2022-05-02 (Actual); Primary Completion 2023-03-02 (Estimated); Study Completion 2023-03-02 (Estimated)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of CB03-154 following single and multiple ascending oral dose administration. | rom the signing of the consent form until 30 days following the last dose of the study drug
  Number of participants with teatment-related adverse events as assessed by CTCAE V5.0 or higher

SECONDARY OUTCOMES:
Maximum Plasma Concentration (Cmax) of CB03-154 | From 1 hour pre-dose to 48 hours post-dose
  Plasma will be collected at multiple timepoints from within 60 minutes pre-dose to 48 hours post-dose
Area Under the Plasma Concentration Versus Time Curve (AUC) of CB03-154 | From 1 hour pre-dose to 48 hours post-dose
  Plasma will be collected at multiple timepoints from within 60 minutes pre-dose to 48 hours post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Frank Lee, M.D, Principal Investigator — Frontage Clinical Services, Inc.
Locations (1):
- Frontage Clinical Services, Inc., Secaucus, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No